CLINICAL TRIAL: NCT05971979
Title: Therapeutic Drug Monitoring - Targeting Improved Effectiveness (TDM-TIME): An Observational Study of Turnaround Time for Therapeutic Drug Monitoring of Antimicrobial Agents in Critically Ill Patients With Respiratory Sepsis
Brief Title: Therapeutic Drug Monitoring - Targeting IMproved Effectiveness
Acronym: TDM-TIME
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B01949
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Pneumonia; Sepsis; Infection, Bacterial
Keywords: drug monitoring; sepsis; antibacterial agents; respiratory tract infections; antimicrobial stewardship
MeSH Terms: conditions — Pneumonia; Sepsis; Bacterial Infections; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients with presumed or confirmed lower respiratory tract infection: Non-interventional. Admitted to intensive care unit. Presumed or confirmed lower respiratory tract infection. Receiving either piperacillin/tazobactam or meropenem. Participants will have samples collected during an antimicrobial dose cycle.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Severe infections can be caused by various organisms, such as bacteria or viruses, and lead to otherwise healthy people getting very unwell, sometimes needing treatment in hospital or even intensive care. For the treatment of bacterial infections to be successful, the correct antibiotics need to be given promptly. Early in the course of illness, clinicians often do not know exactly which bacteria are causing the infection. Furthermore, patients differ in terms of how their bodies process the antibiotics they are given; this means that some may get too much and others too little. This can in turn lead to some patients not being fully cured, and others coming to harm due to side effects of higher doses of these drugs.

For certain types of antibiotics, clinicians are able to measure their levels in the bloodstream, which can help guide dosing. This is called therapeutic drug monitoring, and is commonly used in clinical practice. One of the problems with therapeutic drug monitoring is that it is often not available outside of regular working hours, is costly, and most importantly, provides clinicians with useful information only after a few days of treatment have already been completed. This may be too late to treat these severely ill patients with life-threatening infections, where early and appropriate treatments matter.

The aim of our study, called TDM-TIME, is to look at how long it takes for blood samples to get from the patient to the laboratory to be measured, with the results then communicated back to clinicians. We are further looking to investigate whether steps can be taken to improve these timings, which would lead to shorter times until treatments can be improved. As our study is observational, we will not change anything about the treatment of our patients, but will only be measuring levels of antibiotics in their blood.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Admitted to intensive care;
* Treated for presumed or confirmed lower respiratory tract infection;
* Receiving OR about to receive the first dose of intravenous antimicrobials (either meropenem of piperacillin/tazobactam);
* Valid informed consent OR enrolment through deferred consent appropriate.

Exclusion Criteria:

* Severe anaemia (haemoglobin level < 70 g/L);
* Unlikely to survive 24 hours as judged by the treating physician;
* Study antimicrobial course started more than 24 hours ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria explicitly state otherwise.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Availability of LC-MS/MS results within two dose intervals of antimicrobial (dichotomous) | 48 hours
  Proportion of participants within timeframe for antimicrobial

SECONDARY OUTCOMES:
Time elapsed from peripheral blood collection to LC-MS/MS result availability | 48 hours
  Mean time required for result availability
Time elapsed from first dose of antimicrobial to LC-MS/MS result availability | 72 hours
  Mean time required for result availability from first antimicrobial dose administration
Duration of pre-analytical stage | 24 hours
  Mean time required for pre-analytical stage
Duration of analytical stage | 24 hours
  Mean time required for analytical stage
Duration of post-analytical stage | 24 hours
  Mean time required for post-analytical stage
Therapeutic target attainment (100% fT>4xMIC) | 72 hours
  Proportion of patients attaining target (100% fT>4xMIC)
28-day mortality | 28 days
  Proportion of patients alive at 28 days from enrolment
ICU length of stay | 28 days
  Number of days from ICU admission to discharge
Hospital length of stay | 28 days
  Number of days from hospital admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hansel, MD, Principal Investigator — University of Manchester
Locations (1):
- Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hansel J, Lain J, Erhieyovwe EO, Ismayilli A, Orr J, Keevil BG, Ogungbenro K, Dark PM, Felton TW. A prospective cohort feasibility study of real-time beta-lactam antimicrobial therapeutic drug monitoring in critically ill patients with lower respiratory infection: The TDM-TIME study. J Intensive Care Soc. 2025 Dec 24:17511437251404324. doi: 10.1177/17511437251404324. Online ahead of print. PMID 41459019